CLINICAL TRIAL: NCT03151668
Title: The Effect of Dexmedetomidine on Perfusion Index and Microcirculation in Patients With Severe Sepsis and Septic Shock: Randomized Controlled Study
Brief Title: Effect of Dexmedetomidine on Perfusion Index and Microcirculation in Severe Sepsis and Septic Shock Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Islam Rasmy, Assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: N-14 -2017
Record Dates: First submitted 2017-05-08; First posted 2017-05-12 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Dexmedetomidine

ARMS (2):
- Dexmedetomidin (Experimental)
  Interventions: Drug: Dexmedetomidine
- Midazolam (No Intervention)

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: Dexmedetomidin

SUMMARY:
Septic shock is one of the major causes of death worldwide with in-hospital mortality rates varying between (11.9% to 47.2 %). Alterations in microcirculatory blood flow were associated with high risk of organ dysfunction and death. Experimental studies on septic rats revealed that dexmedetomidine treatment can effectively reduce the generation of inflammatory mediators and yields beneficial effects on endotoxemic animals' microcirculation.

DETAILED DESCRIPTION:
Prospective randomized double blinded study. Investigators planned to enroll (40 cases diagnosed with severe sepsis and/or septic shock ) admitted in 50-bed trauma and surgical ICU Cairo University hospital. Demographic data, cause of ICU admission, source of sepsis, APACHE II score, SOFA score 24 hours after admission. Microcirculatory variables (MFI), peripheral perfusion (PI) and metabolic variables will be measured before drugs administrations and at 2, 4, 6, 24 hours thereafter. The total dose of the infused drugs, The requirement of vasopressor will be evaluated as yes/no and total dose of vasopressor will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* All mechanically ventilated patients who will be clinically suspected of having severe sepsis/septic shock defined by the criteria of the American College of Chest Physicians/ Society of Critical Care Medicine Consensus Conference

Exclusion Criteria:

* Age < 18 years old
* Pregnant patient
* Acute hepatitis or severe liver disease (Child-Pugh class C)
* Left ventricular ejection fraction less than 30%
* Heart rate less than 50 beats/min
* Second or third degree heart block
* Systolic pressure < 90 mmHg despite of infusion of 2 vasopressors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01-04 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of microvascular flow index 6hours after dexmedetomidine infusion | 6 months

SECONDARY OUTCOMES:
The effect of the dexmeditomidine on perfusion index | 6 months
Correlation between perfusion index and microvascular flow index in septic shock patients | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo, Egypt

REFERENCES:
- [Background] Rasmy I, Mohamed H, Nabil N, Abdalah S, Hasanin A, Eladawy A, Ahmed M, Mukhtar A. Evaluation of Perfusion Index as a Predictor of Vasopressor Requirement in Patients with Severe Sepsis. Shock. 2015 Dec;44(6):554-9. doi: 10.1097/SHK.0000000000000481. PMID 26529657
- [Background] Zhang J, Wang Z, Wang Y, Zhou G, Li H. The effect of dexmedetomidine on inflammatory response of septic rats. BMC Anesthesiol. 2015 May 1;15:68. doi: 10.1186/s12871-015-0042-8. PMID 25929655
- [Background] Miranda ML, Balarini MM, Bouskela E. Dexmedetomidine attenuates the microcirculatory derangements evoked by experimental sepsis. Anesthesiology. 2015 Mar;122(3):619-30. doi: 10.1097/ALN.0000000000000491. PMID 25313879